CLINICAL TRIAL: NCT04310423
Title: An Inflammatory Challenge Using Endotoxin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lara Ray, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 19-001561
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder; Inflammatory Response; Craving; Depressed Mood
MeSH Terms: conditions — Alcoholism; Consciousness Disorders | interventions — Sodium Chloride; Endotoxins

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, placebo-controlled, parallel-group study of low dose endotoxin (0.8 ng/kg)
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study team, medical personnel, and participants will be blind to drug condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Matched to endotoxin
  Interventions: Drug: Placebo
- Endotoxin (Experimental): Bolus dose of endotoxin (0.8 ng/kg)
  Interventions: Biological: Endotoxin

INTERVENTIONS:
Drug: Placebo — Matched to endotoxin
  Other Names: Saline (0.9%)
  Arms: Placebo
Biological: Endotoxin — Bolus dose of 0.8 ng/kg
  Other Names: Escherichia coli
  Arms: Endotoxin

SUMMARY:
The study design consists of a randomized, double-blind, placebo-controlled trial of low dose endotoxin. The low dose endotoxin challenge induces a transient systemic inflammatory response with normalization of cytokine levels within hours. This "phasic" inflammation is distinct from chronic ("tonic") levels of inflammation that may be present with AUD. A total of 38 non-treatment seeking heavy drinking men and women and 38 light drinking healthy controls will participate in the study. Recruitment will be monitored to ensure the two groups are matched by gender. Eligible participants will be randomly assigned, stratified by gender and BDI-II severity, to receive a single I.V. infusion of either low dose endotoxin (0.8 ng/kg of body weight) or placebo (same volume of 0.9% saline solution) at the UCLA Outpatient Clinical and Translational Research Center (CTRC). All participants will complete an alcohol cue-exposure paradigm and reward responsiveness assessment 2 hours post infusion, which is the time of expected peak cytokine response. All participants will also complete an fMRI alcohol cue-reactivity paradigm at 3 hours post infusion. Plasma levels of proinflammatory cytokines [i.e., Interleukin-6 (IL-6) and tumor necrosis factor-α (TNF- α)], mood, and alcohol craving, will be assessed at baseline and then hourly for four hours post infusion.

DETAILED DESCRIPTION:
RECRUITMENT: Participants will be recruited from the community through online and newspaper advertisements. Campaigns in local buses and print publications (e.g., LA Weekly) will also be implemented. Targeted recruitment will also take place through a lab database of previous study participants who agreed to be contacted for future studies.

TELEPHONE SCREEN: Individuals who call the lab (in response to flyers and advertisements) expressing interest in the study will receive detailed information about the study procedures, and if they remain interested they will complete a telephone screen performed by a trained research assistant for self-reported inclusion and exclusion criteria. Those who appear eligible will be invited to the laboratory for an initial in-person screening session.

INITIAL SCREENING: Prior to conducting any research related procedures, research staff will conduct the informed consent process, which details the procedures to take place during the screening visit. Informed consent will be a three part process. First, participants will be asked to read and provide verbal consent for breathalyzer. If the breathalyzer is above 0.000, the visit will be stopped and the participant will not be compensated. The participant will be given an opportunity to reschedule the visit for another day. If the breathalyzer test is negative, the written informed consent form will be reviewed and signed by the participant and study staff outlining procedures for the initial screening visit. A second written consent form will be reviewed and signed in the presence of the study physician at the medical screening visit if the participant is found eligible to continue to that visit. At the initial screening visit, subjects will be asked to provide a urine sample to test for drugs of abuse and pregnancy (if female), and will complete a series of individual differences measures (described in detail below). This visit should take approximately 2 hours. Following the initial in-person screening, the study coordinator will meet with the PI to determine if the participant is eligible to continue to the medical screening based on study inclusion/exclusion criteria.

MEDICAL SCREENING: Those participants who appear to be eligible after the initial screening visit, will then be scheduled for a second screening visit. This visit will be conducted by the study physician and will start with a breathalyzer test. If the breathalyzer is above 0.000, the visit will be stopped and the participant will not be compensated. The participant will be given an opportunity to reschedule the visit for another day. If the breathalyzer test is negative, the physician will conduct the second written (experimental) consent; medical history interview and physical exam. In addition, a urine drug screen test will be repeated. The participant will then be accompanied by research personnel to the CTRC for blood specimen collection including Comprehensive Metabolic Panel and Complete Blood Count to evaluate overall health; and EKG to screen for medical conditions that could make study participation medically unsafe. The study physician will review each participant's medical history, vital signs, weight, review of systems, and laboratory tests, including liver function tests (LFTs), drug screen, chemistry screen, and urine pregnancy screen to determine if it is medically safe for the participant to take the study medication. Any subject who is excluded from the study will be compensated for their time in the screening session and will be offered referrals for alcohol treatment in the community.

RANDOMIZATION/INFLAMMATORY CHALLENGE: Upon arrival to the CTRC, eligibility for the inflammatory challenge will be reviewed to ensure that none of the exclusion criteria have been met as described above. A nurse, who will be blind to the condition, will insert a catheter with a heparin lock into the non-dominant forearm for drug administration and hourly blood draws. Each participant will be randomly assigned to receive either low-dose endotoxin (0.8 ng/kg of body weight administered) or placebo (same volume of 0.9% saline), which will be administered by the nurse as an intravenous bolus. The endotoxin will be derived from Escherichia coli (E. Coli group O:113: BB-IND 12948 to M.R.I) and will be provided by the National Institutes of Health Clinical Center as a reference endotoxin for studies of experimental inflammation in humans. Participants will complete assessments as outlined below at baseline and every hour for 4 hours post-infusion. One standard meal and one snack will be provided by the CTRC to each participant during the experimental visit. At the end of the experimental period, participants will have the catheter removed and will be discharged with instructions to abstain from consuming alcohol for 24 hours after discharge. A follow-up phone call by the study physician will be conducted the day after the inflammatory challenge and again 1-2 weeks later to assess for any adverse events.

The study physician (Dr. Miotto) will be on-call and will manage any adverse events during the inflammatory challenge. She will consult with Dr. Irwin, Co-I, as needed to manage adverse events. In the event that significant medical problems are encountered, the blind will be broken and appropriate medical treatment will be provided. Individuals who meet the following stopping criteria will discontinue study-related data collection procedures (cytokine assays and cue exposure paradigm):

1. >1 SAE at least possibly related to endotoxin administration
2. >2 Grade 3 (severe) adverse events at least possibly related to endotoxin administration, based on the FDA Guidance Document "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" ALCOHOL CUE REACTIVITY SESSION (CR): Approximately 2 hours after receiving intravenous endotoxin (or matched placebo), participants will complete the cue-exposure paradigm. Alcohol cue exposure will follow well-established experimental procedures. Sessions will begin with a 3-minute relaxation period. Participants will then hold and smell a glass of water for 3 minutes to control for the effects of simple exposure to any potable liquid. Next, participants will hold and smell a glass of their preferred alcoholic beverage for 3 minutes. Order is not counterbalanced because of carryover effects that are known to occur. Participants (who are smokers) will be allowed a smoke break immediately prior to and immediately after the CR assessment. After every 3 minute period, participants will rate their urge to drink on the Alcohol Urge Questionnaire.

REWARD RESPONSIVENESS: Approximately 2 hours after receiving intravenous endotoxin (or matched placebo), participants will complete the reward responsiveness paradigm, including the Probabilistic Reward Task (PRT) and Reward Responsiveness Scale (RRS). The PRT is a 25-minute task that will be administered at baseline and hour 2. The task assesses behavioral modulation as a function of reward-based reinforcement (i.e. reward seeking) by asking participants to respond to stimuli, eliciting a response bias by introducing an asymmetric reinforcer ratio. The RRS is a self-report questionnaire that measures reward responsiveness by asking subjects to rate their agreement with various statements on a 4-point Likert scale.

NEUROIMAGING CUE-REACTIVITY (fMRI): Approximately 3 hours after receiving intravenous endotoxin (or matched placebo), participants will complete a functional magnetic resonance imaging (fMRI) scan. This scan will include an fMRI visual alcohol cue-reactivity paradigm, which will follow well-established procedures. The alcohol cues task consists of viewing visual alcohol, negative, and neutral cues, presented in six 120-s epochs (total scan duration: 12 minutes), with each epoch consisting of four 24-s blocks (one block of alcohol cues, one block of neutral cues, one block of negative images, and one block of fixation). Alcohol blocks will be specific to beverage type (beer, wine, or liquor), with two blocks of each beverage type. Prior to scanning, participants will rate their craving on a four-point scale and will also provide ratings of their craving immediately following each cue block.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 21 and 45
2. Be non-treatment seeking for AUD
3. Have had at least one alcoholic beverage in the last 30 days
4. FOR HEAVY DRINKERS: Alcohol Use Disorder Identification Test (AUDIT) score between 8 - 15; FOR LIGHT DRINKERS: AUDIT score < 4
5. FOR HEAVY DRINKERS: Report drinking at binge levels at least 1 time in the past month (5+ drinks/day for men, 4+ drinks/day for women); FOR LIGHT DRINKERS: report no occasions of binge drinking in the past month

Exclusion Criteria:

1. Have a current (last 12 months) DSM-5 diagnosis of substance use disorder for any psychoactive substances other than alcohol and nicotine
2. Have a lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder
3. Have current moderate to severe depression as indicated by a score of ≥ 21 on the Beck Depression Inventory - II (BDI-II)
4. Have current suicidal ideation or lifetime history of suicide attempt as reported on the Columbia-Suicide Severity Rating Scale (C-SSRS)
5. Have a positive urine screen for drugs other than cannabis;
6. Have clinically significant alcohol withdrawal symptoms as indicated by a score ≥ 8 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-R)
7. Have an intense fear of needles or have had any adverse reactions to needle puncture
8. Be pregnant, nursing, or planning to become pregnant while taking part in the study; and must agree to one of the following methods of birth control (if female), unless she or partner are surgically sterile:

   * Oral contraceptives
   * Contraceptive sponge
   * Patch
   * Double barrier
   * Intrauterine contraceptive device
   * Etonogestrel implant
   * Medroxyprogesterone acetate contraceptive injection
   * Complete abstinence from sexual intercourse
   * Hormonal vaginal contraceptive ring
9. Have a medical condition that may interfere with safe study participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes, autoimmune or inflammatory disease)
10. Have clinically significant abnormal EKG
11. Have > Grade 2 laboratory abnormalities, based on FDA Guidance Document "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials"
12. Have any other circumstances that, in the opinion of the investigators, compromises participant safety
13. Have non-removable ferromagnetic objects in body
14. Have claustrophobia
15. Have serious head injury or prolonged period of unconsciousness (>30 minutes)

Exclusionary Criteria for Inflammatory Challenge Visits:

1. BrAC > 0.000 g/dl
2. clinical withdrawal (CIWA-R) score ≥ 8
3. blood pressure ≤ 90/60 or ≥ 160/120
4. resting pulse ≤ 50 beats/minute or > 100 beats/minute
5. temperature ≥ 99.5°F
6. recent (past 2 weeks) acute illness or vaccination
7. score of 10+ on Physical Sickness Symptoms Assessment

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Addictions Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening procedures for participants were conducted from 2021 - 2023; therefore, given the COVID-19 pandemic, initial screening procedures were conducted via HIPAA-compliant telemedicine software. Following, participants completed a medical screening visit at the Clinical and Translational Research Center (CTRC) at UCLA. Following, participants completed the experimental visit at the CTRC and the UCLA Center for Cognitive Neuroscience (CCN).
Pre-assignment Details: Participants completed an initial and medical screening visit for eligibility prior to the randomization assignment.
Period: Overall Study
Arm/Group | Placebo | Endotoxin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Endotoxin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.80 (7.58) | 30.30 (6.53) | 29.05 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Alcohol Use Disorder Identification Test [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorder Identification Test (AUDIT) is a 10-item self-report measure of severity of alcohol use. AUDIT total sum score can range from 0-40, with higher scores indicating higher alcohol use severity.
  units on a scale | 12.00 (2.66) | 13.30 (6.18) | 12.65 (4.68)
Beck Depression Inventory - 2 [Mean (Standard Deviation); unit: score on a scale] — The Beck Depression Inventory - 2 (BDI-II) is a 21-item self-report questionnaire of depressive symptoms. BDI-2 total sum score can range from 0-63, with higher scores indicative of more depressive symptoms.
  score on a scale | 7.40 (6.28) | 7.80 (7.90) | 7.60 (6.95)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.99 (4.07) | 27.25 (3.72) | 26.12 (3.97)
Drinks per Drinking Day [Mean (Standard Deviation); unit: drinks/drinking day] — Drinks per drinking day (DPDD) was calculated based off of Timeline Follow Back (TLFB) interview in which participants reported their alcohol use over the past 30 days. DPDD was calculated as the average drinks consumed on drinking days.
  drinks/drinking day | 4.58 (1.95) | 4.12 (1.40) | 4.35 (1.67)
Structured Clinical Interview for DSM-5 Alcohol Use Disorder Symptoms [Mean (Standard Deviation); unit: symptoms] — Past 12-month Alcohol Use Disorder (AUD) total symptom score was assessed by clinician-administered Structured Clinical Interview for DSM-5 (SCID). The SCID is a semi-structured interview designed for the diagnosis of psychiatric disorders, including AUD. The Alcohol Use Disorder module assessed 11 symptoms of AUD, with 2 or more symptoms endorsed indicating the presence of AUD. The total symptoms could range from 0-11, with a higher score indicating more symptoms of AUD.
  symptoms | 4.20 (1.93) | 4.10 (1.85) | 4.15 (1.84)
Reward Relief Habit Drinking Scale [Count of Participants; unit: Participants] — The Reward, Relief, Habit Drinking Scale (RRHDS) is a four-item self-report questionnaire. The first question asked participants their primary reason for drinking alcohol (i.e. reward, relief or habit) while the remaining three questions use a 1-7 scale to rate how often they drank alcohol for its rewarding effects, relieving effects, or our of habit, with higher ratings indicating drinking more often for the specified reason. Participants were classified into reward, relief and habit drinking sub-types based on the highest rating provided for questions 2-4.
  Participants
    Reward | 9 | 9 | 18
    Relief | 1 | 1 | 2
    Habit | 0 | 0 | 0
Years of Education [Mean (Standard Deviation); unit: years] | 16.00 (2.45) | 16.90 (2.13) | 16.45 (2.28)

OUTCOME MEASURES:

1. Primary Outcome: Cue-induced Craving
Description: Alcohol Urge Questionnaire (AUQ) score is the primary outcome for the cue-reactivity paradigm. The AUQ is comprised of eight items rated on a 7-point Likert scale with items related to the subjective experience of alcohol craving. The minimum value is 8 and the maximum value is 56 with a higher score indicating greater subjective alcohol craving. Phasic craving for alcohol following alcohol cue exposure was assessed using the first and last items from the AUQ during an alcohol cue reactivity paradigm at baseline and at time of expected peak cytokine response (T2). This subscale of 2 items about desire to drink rated on a 7-point Likert scale provided a minimum possible value of 2 and a maximum value of 14, with higher values indicating a higher craving to drink alcohol. The investigators are primarily interested in whether low dose endotoxin increases cue-induced craving for alcohol in non-treatment-seeking heavy drinkers, relative to placebo.
Time Frame: The cue-reactivity paradigm is conducted at baseline and at 2 hours post-infusion of placebo or low dose endotoxin during the experimental visit.
Population: All randomized participants included in analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Endotoxin
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 4.5004 (0.9622) | 7.9081 (0.9604)
  Two Hours Post-Baseline: number analyzed (Participants) | 10 | 9
  Two Hours Post-Baseline | 4.5004 (0.9622) | 5.6178 (0.9858)
Statistical Analysis 1: Comparison: Placebo vs Endotoxin; Treatment x Time interaction for alcohol cue-induced alcohol craving; Test type: Other; p = 0.036, Mixed Models Analysis

2. Primary Outcome: Change in Negative Mood
Description: The Profile of Mood States (POMS) is a self-report questionnaire that measures dimensions of mood. Four items from the POMS were summed to calculate the negative mood subscale. The items included "discouraged," downhearted," "uneasy," and "anxious." Participants rated the extent that they felt items "right now" on a scale from 0-4, with higher scores indicating more endorsement of the items. Items were summed to calculate negative mood subscale with the score ranging from 0-16, with higher scores indicating higher negative mood. The investigators were interested in whether low dose endotoxin would increase negative mood as compared to placebo.
Time Frame: The POMS will be completed at 5 timepoints during the experimental visit. Specifically, negative mood will be assessed at baseline (prior to infusion) and 1 hour, 2 hours, 3 hours, and 4 hours post-infusion of placebo or low dose endotoxin.
Population: All participants were included in the analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Endotoxin
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 0.60 (0.27) | 0.80 (0.36)
  One Hour Post-Baseline | 0.50 (0.34) | 0.90 (0.43)
  Two Hours Post-Baseline: number analyzed (Participants) | 10 | 9
  Two Hours Post-Baseline | 0.50 (0.27) | 0.90 (0.31)
  Three Hours Post-Baseline | 1.70 (0.88) | 1.70 (0.72)
  Four Hours Post-Baseline | 0.90 (0.53) | 1.70 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Endotoxin; Two-way Treatment x Time interaction; Test type: Other; p > 0.05, Mixed Models Analysis

3. Secondary Outcome: Change in Reward Responsiveness
Description: The Reward Responsiveness Scale (RRS) measures self-report reward responsiveness. The RRS scale consists of 8 items on a 4-point scale, with the sum total score of items ranging from 8-32, where higher scores indicate higher reward responsiveness. The measure was completed electronically. The investigators are interested in whether low dose endotoxin will decrease reward responsiveness as compared to placebo.
Time Frame: The RRS will be completed at 2 timepoints during the experimental visit. Specifically, reward responsiveness will be assessed at baseline (prior to infusion) and 2 hours post-infusion of placebo or low dose endotoxin.
Population: All participants included in analysis; participants completed RRS at baseline and two-hours post-baseline (T2).
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Endotoxin
Number analyzed (Participants) | 10 | 10
scores on scale
  RRS Baseline | 25.60 (1.11) | 26.20 (0.98)
  RRS Two Hours Post-Baseline | 25.50 (1.27) | 26.22 (1.24)
Statistical Analysis 1: Comparison: Placebo vs Endotoxin; Treatment x Time interactions; Test type: Other; p > 0.05, Mixed Models Analysis

4. Secondary Outcome: Change in Reward Responsiveness
Description: The Probabilistic Reward Task (PRT) is a signal detection learning task that assesses reward learning from which two subscales were derived: logd is a measure of discriminability, or how difficult it is for the subjects to discriminate between the signals, while logb is a measure of response bias, or subjects' preference for the response paired with the more frequent reward. Higher logd values indicate a better ability to discriminate between reward signals (logd=1⁄2 log(Richcorrect*Leancorrect)/(Richincorrect*Leanincorrect)). Higher logb values indicate better reward sensitivity (logb=1⁄2 log(Richcorrect*Leanincorrect)/(Richincorrect*Leancorrect)). The range of possible logb and logd subscale values is between -2.48 to 2.48. The measure was completed electronically. The investigators are interested in whether low dose endotoxin will decrease reward responsiveness as compared to placebo.
Time Frame: The PRT will be completed at 2 timepoints during the experimental visit. Specifically, reward responsiveness will be assessed at baseline (prior to infusion) and 2 hours post-infusion of placebo or low dose endotoxin.
Population: All participants included in analysis; participants completed PRT at baseline and two-hours post-baseline (T2).
Measure: Mean (Standard Error); unit: scores on task
Arm/Group | Placebo | Endotoxin
Number analyzed (Participants) | 10 | 10
scores on task
  PRT logd Baseline | 1.46 (0.13) | 1.29 (0.16)
  PRT logd Two Hours Post-Basleine | 1.98 (0.33) | 1.27 (0.16)
  PRT logb Baseline | -0.07 (0.03) | 0.16 (0.05)
  PRT logb Two Hours Post-Baseline | 0.31 (0.38) | 0.20 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Endotoxin; Treatment x Time interactions; Test type: Other; p > 0.05, Mixed Models Analysis

5. Secondary Outcome: Effect on Neural Alcohol Cue-reactivity
Description: The fMRI scan will include a cue-reactivity paradigm in which participants will view images of alcoholic beverages, non-alcoholic beverages, negative images, and fixation cross. Participants will be asked to rate their alcohol craving before the scan and after each cue block. The investigators are interested in determining the effects of endotoxin on neural alcohol cue-reactivity. An alcohol beverage > non-alcohol beverage contrast was specified in the first-level model for each subject, and FSL's FLAME 1 was used to conduct group-level analyses (endotoxin vs. placebo) to identify significant brain clusters in which individuals who received placebo had greater activation for alcohol beverages compared to non-alcohol beverages than those who received endotoxin. Outcome measure below indicates the voxel size of said significant clusters.
Time Frame: The fMRI scan will be completed during the experimental visit. Specifically, participants will undergo the neuroimaging scan at 3 hours post-infusion of placebo or low dose endotoxin.
Population: All participants included in analysis. The outcome measure data below indicates the voxel size of significant clusters identified in which individuals who received placebo had greater activation for alcohol beverages compared to non-alcohol beverages than those who received endotoxin. Therefore, only one Arm/Group is reported, as the neuroimaging analyses used FSL software wherein the outcome is the identification of these significant clusters.
Measure: Number; unit: Voxels
Groups:
- Placebo > Endotoxin (Alcohol vs. Beverage Cues) at T3: Placebo matched to endotoxin>Bolus dose of endotoxin (0.8 ng/kg)
  Placebo: Matched to endotoxin
Arm/Group | Placebo > Endotoxin (Alcohol vs. Beverage Cues) at T3
Number analyzed (Participants) | 20
Voxels
  Left Postcentral Gyrus Significant Cluster | 3190
  Right Thalamus Significant Cluster | 1942
  Left Inferior Temporal Gyrus Cluster | 931
  Left/Right Precuneus Cluster | 920
  Right Precentral Gyrus | 518
Statistical Analysis 1: Comparison: Placebo > Endotoxin (Alcohol vs. Beverage Cues) at T3; Main effect of treatment on alcohol cue-elicited brain activation; Test type: Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study duration from 2021-2023.
Description: Adverse event information was collected during 4-hour inflammatory challenge and then for one week following the challenge. FDA Guidance Document "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" was used to inform adverse events. Stopping criteria was met if there was emergence of an SAE or more than 1 Grade 3 (severe) adverse event at least possibly related to endotoxin.
Arm/Group | Placebo | Endotoxin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Endotoxin (N=10)
Fever (Immune system disorders) | 0 (0) | 2 (2)
Nausea (Immune system disorders) | 0 (0) | 4 (4)
Shivering (Immune system disorders) | 0 (0) | 7 (7)
Fatigue (Immune system disorders) | 5 (5) | 7 (7)
Shortness of Breath (Immune system disorders) | 0 (0) | 2 (2)
Muscle Pain (Immune system disorders) | 1 (2) | 4 (4)
Arm Rash (Immune system disorders) | 0 (0) | 1 (1)
Hypertension (Immune system disorders) | 0 (0) | 1 (1)
Headache (Immune system disorders) | 2 (2) | 2 (2)
Lightheadedness (Immune system disorders) | 0 (0) | 1 (1)
Low Back Pain (Immune system disorders) | 0 (0) | 1 (1)
Injection Site Pain (Immune system disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to COVID-19 pandemic-related research delays in 2020, as well as a FDA clinical hold on Endotoxin product testing and release, the original target of 38 heavy drinking participants and 38 light-drinking controls was not met. The study team was able to randomize a total of 20 heavy drinking participants and leveraged 20 light-drinking matched control participants from sub-investigator Dr. Naomi Eisenberger's previously completed Endotoxin study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT04310423/Prot_SAP_001.pdf